CLINICAL TRIAL: NCT02557308
Title: An Observational, Prospective, Cohort Study to Evaluate Safety and Efficacy of Remsima™ in Patients With Ankylosing Spondylitis
Brief Title: An Observational Study to Evaluate Safety and Efficacy of Remsima™ in Patients With Ankylosing Spondylitis
Status: Terminated | Type: Observational
Why Stopped: Terminated
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Other Study IDs: CT-P13 4.4
Record Dates: First submitted 2015-05-15; First posted 2015-09-23 (Estimated); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Remsima™: Patients who have received only Remsima were included in this analysis group
- Switch to Remsima I: Patients who switched from Remicade to Remsima were included in this analysis group.
- Switch to Remsima II: Patients who switched to Remsima from biologic treatment other than Remicade were included in this analysis group
- Remicade: Patients who switched from Remsima to Remicade were included in this analysis group.
- Switch to Remicade I: Patients who switched from Remsima to Remicade were included in this analysis group.
- Switch to Remicade II: Patients who switched to Remicade from biologic treatment other than Remsima were included in this analysis group.
- Other anti-TNF drugs: Following patients were included in other anti-TNF group.
  * Patients who have received only anti-TNF other than Remsima or Remicade
  * Patients who switched from biologic treatment other than anti-TNF before study enrollment to anti-TNF other than Remsima or Remicade
- Switch to Other Anti-TNF: Patients who switched from Remsima or Remicade to other anti-TNF other than Remicade were included in this analysis group

SUMMARY:
An Observational, Prospective Cohort Study to Evaluate Safety and Efficacy of RemsimaTM in Patients with Ankylosing Spondylitis

DETAILED DESCRIPTION:
This is a longitudinal, observational, prospective cohort study to assess the safety and efficacy of RemsimaTM in patients with AS in comparison with patients receiving other TNF blockers. For the RemsimaTM cohort data will be collected for patients who commence treatment with RemsimaTM in accordance with the product label at the time of enrolment. Patients who have been treated with Remicade® prior to enrolment, their dosing schedule will be continued appropriately. This observational study allows drug switching between anti-TNF drugs. If switched to RemsimaTM, data will be collected until the end of study for each patient. If switched to other anti-TNF drugs (infliximab (Remicade®), etanercept, adalimumab and etc.), data will be collected until 1 year from the day of switch or until the end of study for each patient, whichever reaches earlier. For switched patients, their assessment schedule will be re-started from the day of switch. Patients will undergo safety and efficacy assessments in accordance with routine medical practice. The decision to treat with RemsimaTM will be independent of the decision to enroll the patient in this registry.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Patients with active AS
* Patients who meet the following conditions can be enrolled:

  i) The RemsimaTM cohort will include all patients who will start RemsimaTM at the time of enrolment in accordance to the approved product label ii) Patients who have started to be treated with an established anti -TNF such as Infliximab (Remicade®), Etanercept, Adalimumab and etc. within 6 months
* Female patients of childbearing potential who agree to use of adequate contraception to prevent pregnancy and continuation of contraceptive use for at least 6 months after their final dose of RemsimaTM.
* Patients (or legal guardian, if applicable) who are willing to give informed consent for long term follow-up including access to all medical records

Exclusion Criteria:

* Patients with a history of hypersensitivity to infliximab
* Patients with a current or past history of chronic infection
* Current diagnosis of TB or severe or chronic infections (e.g. sepsis, abscess or opportunistic infections or invasive fungal infections), or a past diagnosis of TB or severe or chronic infection, without sufficient documentation of complete resolution following treatment.
* Recent exposure to persons with active TB, or a positive test result for latent TB (defined as a positive interferon-γ release assay [IGRA] with a negative examination of chest X-ray) at Screening.
* Patients with moderate or severe heart failure (NYHA class III/IV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 1000 male or female patients with confirmed diagnosis of AS.
Sampling Method: Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2015-05-26 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klara Sirova, Principal Investigator — Revmatologie MUDr. Klara Sirova s.r.o. Chelčického 616/12 , 702 00, Czech Republic

REFERENCES:
- [Derived] Cheon JH, Nah S, Kang HW, Lim YJ, Lee SH, Lee SJ, Kim SH, Jung NH, Park JE, Lee YJ, Jeon DB, Lee YM, Kim JM, Park SH. Infliximab Biosimilar CT-P13 Observational Studies for Rheumatoid Arthritis, Inflammatory Bowel Diseases, and Ankylosing Spondylitis: Pooled Analysis of Long-Term Safety and Effectiveness. Adv Ther. 2021 Aug;38(8):4366-4387. doi: 10.1007/s12325-021-01834-3. Epub 2021 Jul 12. PMID 34250583

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant flow was summarized by all analysis groups as prespecified in Statistical Analysis Plan.
Pre-assignment Details: A total of 350 patients were screened, and 329 patients were enrolled.
Groups:
- Remsima: Patients who have received only Remsima were included in this analysis group
- Switch to Remsima: Patients who switched from Remicade to Remsima were included in this analysis group.
- Switch to Remsima II: Patients who switched to Remsima from biologic treatment other than Remicade will be included in this analysis group.
- Remicade: Patients who have received only Remicade were included in this analysis group.
- Switch to Remicade: Patients who switched from Remsima to Remicade were included in this analysis group.
- Switch to Remicade II: Patients who switched to Remicade from biologic treatment other than Remsima will be included in this analysis group.
- Other Anti-TNF: Following patients were included in other anti-TNF group.
  * Patients who have received only anti-TNF other than Remsima or Remicade
  * Patients who switched from biologic treatment other than anti-TNF before study enrolment to anti-TNF other than Remsima or Remicade
- Switch to Other Anti-TNF: Patients who switched from Remsima or Remicade to other anti-TNF other than Remicade will be included in this analysis group.
Period: Overall Study
Arm/Group | Remsima | Switch to Remsima | Switch to Remsima II | Remicade | Switch to Remicade | Switch to Remicade II | Other Anti-TNF | Switch to Other Anti-TNF
Started | 124 | 23 | 10 | 3 | 5 | 0 | 146 | 18
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not Completed | 124 | 23 | 10 | 3 | 5 | 0 | 146 | 17
Not completed — Withdrawal by Subject | 11 | 3 | 2 | 0 | 1 | 0 | 10 | 1
Not completed — Disease Progression | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 4 | 1 | 2 | 0 | 0 | 0 | 4 | 1
Not completed — Lost to Follow-up | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study Close | 98 | 18 | 5 | 3 | 1 | 0 | 123 | 5
Not completed — Except for study close | 5 | 0 | 0 | 0 | 3 | 0 | 6 | 10

BASELINE CHARACTERISTICS:
Population: All patients data were analyzed; however, there were 0 patients recruited in the "Switch to Remicade II" groups.
Groups:
- Other Anti-TNF Drugs: Following patients were included in other anti-TNF group.
  * Patients who have received only anti-TNF other than Remsima or Remicade
  * Patients who switched from biologic treatment other than anti-TNF before study enrolment to anti-TNF other than Remsima or Remicade
- Total: Total of all reporting groups
Arm/Group | Remsima | Switch to Remsima I | Switch to Remsima II | Remicade | Switch to Remicade I | Switch to Remicade II | Other Anti-TNF Drugs | Switch to Other Anti-TNF | Total
Number analyzed (Participants) | 124 | 23 | 10 | 3 | 5 | 0 | 146 | 18 | 329
Age, Continuous [Median (Full Range); unit: years] | 37.0 [18 to 75] | 42.0 [22 to 59] | 46.0 [24 to 78] | 32.0 [30 to 57] | 41.0 [29 to 62] |  | 38 [18 to 80] | 39 [20 to 64] | 38.0 [18 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 3 | 3 | 1 | 2 | 0 | 26 | 5 | 66
  Male | 98 | 20 | 7 | 2 | 3 | 0 | 120 | 13 | 263
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 97 | 23 | 3 | 3 | 5 | 0 | 129 | 8 | 268
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 27 | 0 | 7 | 0 | 0 | 0 | 17 | 10 | 61
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Number and Percentage of Patients With the Following Adverse of Events of Special Interest (ESI)
Description: * Hepatitis B virus reactivation
  * Congestive heart failure
  * Opportunistic infections (excluding tuberculosis)
  * Serious infections including sepsis (excluding opportunistic infections and tuberculosis)
  * Tuberculosis (TB)
  * Serum sickness (delayed hypersensitivity reactions)
  * Haematological reactions
  * Systemic lupus erythematosus/lupus-like syndrome
  * Demyelinating disorders
  * Lymphoma (not hepatosplenic T cell lymphoma)
  * Hepatobiliary events
  * Hepatosplenic T cell lymphoma (HSTCL)
  * Serious infusion reactions during a re-induction regimen following disease flare
  * Sarcoidosis/sarcoid-like reactions
  * Leukaemia
  * Malignancy (excluding lymphoma)
  * Skin cancer
  * Pregnancy exposure
  * Infusion related reaction (IRR)/hypersensitivity/anaphylactic reaction
Time Frame: Duration of study participation (up to 5 years)
Population: All patients data were analyzed; however, there were 0 patients recruited in the "Switch to Remicade II" groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Remsima | Switch to Remsima I | Switch to Remsima II | Remicade | Switch to Remicade I | Switch to Remicade II | Other Anti-TNF | Switch to Other Anti-TNF
Number analyzed (Participants) | 124 | 23 | 10 | 3 | 5 | 0 | 146 | 18
Participants
  TEAE of congestive heart failure | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TEAE of Opportunistic infections (excluding tuberculosis) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TEAE of Serious infections including sepsis (excluding opportunistic infections and tuberculosis) | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  TEAE of tuberculosis | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  TEAE of Haematological reactions | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1
  TEAE of Hepatobiliary events | 9 | 1 | 2 | 0 | 0 | 0 | 9 | 0
  TEAE of Malignancies (excluding lymphoma) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  TEAE of Infusion related reaction/hypersensitivity/ anaphylactic reaction | 3 | 0 | 0 | 1 | 1 | 0 | 2 | 1

2. Secondary Outcome: The Number and Percentage of Patients Achieving BASDAI 50
Description: Efficacy was assessed by the evaluation of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI). The BASDAI questionnaire consists of 6 component questions about the disease activity. For each question the possible answer from the patient is a whole number from 0 to 10 inclusive where 0 = None and 10 = Very severe. The BASDAI score is generated from the set of 6 questions and calculated using the following formula BASDAI = [Q1+Q2+Q3+Q4+([Q5+Q6]/2)]/5. The number and percentage of patients achieving BASDAI 50 will be displayed. BASDAI 50 is defined as a 50% decrease of the baseline BASDAI score. Percentages will be calculated using the number of patients who perform the assessment at each time point.
Time Frame: Month 6 ~ Month 48 (every 6 months ± 6 weeks)
Population: Efficacy analysis was only performed in the Remsima, Switch to Remsima, Remicade and Switch to Remicade analysis groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Remsima | Switch to Remsima | Remicade | Switch to Remicade
Number analyzed (Participants) | 98 | 20 | 3 | 4
Participants
  Month 6: number analyzed (Participants) | 85 | 16 | 3 | 4
  Month 6 | 60 | 5 | 3 | 2
  Month 12: number analyzed (Participants) | 56 | 14 | 1 | 2
  Month 12 | 35 | 1 | 1 | 1
  Month 18: number analyzed (Participants) | 27 | 0 | 1 | 0
  Month 18 | 16 | 0 | 1 | 0
  Month 24: number analyzed (Participants) | 16 | 0 | 0 | 0
  Month 24 | 13 | 0 | 0 | 0
  Month 30: number analyzed (Participants) | 13 | 0 | 0 | 0
  Month 30 | 11 | 0 | 0 | 0
  Month 36: number analyzed (Participants) | 14 | 0 | 0 | 0
  Month 36 | 12 | 0 | 0 | 0
  Month 42: number analyzed (Participants) | 0 | 0 | 0 | 0
  Month 42 | 0 | 0 | 0 | 0
  Month 48: number analyzed (Participants) | 6 | 0 | 0 | 0
  Month 48 | 6 | 0 | 0 | 0

3. Secondary Outcome: Descriptive Statistics for BASFI
Description: The Bath Ankylosing Spondylitis Functional Index (BASFI) questionnaire consists of 10 component questions measuring functionality. Each item was given a rating by the patient which is a whole number from 0 to 10 inclusive where 0 = Easy and 10 = Impossible. The BASFI score is generated from the mean of the scores for the 10 items. The lowest score is 0 and the highest score is 10, with higher scores indicating a higher degree of functional limitation in patients.
Time Frame: Day 0 ~ Month 48 (every 6 months ± 6 weeks)
Population: The Efficacy Analysis set consisted of all patients who received at least one infliximab dose (Remsima or Remicade) and providing at least one post treatment efficacy result during the analysis period. Efficacy analysis was only performed in the Remsima, Switch to Remsima, Remicade and Switch to Remicade analysis groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Remsima™ | Switch to Remsima | Remicade | Switch to Remicade
Number analyzed (Participants) | 98 | 20 | 3 | 4
score on a scale
  Day 0: number analyzed (Participants) | 97 | 20 | 3 | 4
  Day 0 | 4.10 (2.684) | 1.35 (1.746) | 2.07 (3.239) | 1.65 (2.014)
  Month 6: number analyzed (Participants) | 86 | 16 | 3 | 4
  Month 6 | 1.38 (1.498) | 1.10 (1.614) | 0.70 (1.212) | 1.93 (1.427)
  Month 12: number analyzed (Participants) | 56 | 14 | 1 | 2
  Month 12 | 1.36 (1.553) | 1.43 (1.679) | 3 | 3.05 (1.061)
  Month 18: number analyzed (Participants) | 28 | 2 | 1 | 0
  Month 18 | 1.38 (1.774) | 1.70 (2.121) | 2.40 |
  Month 24: number analyzed (Participants) | 17 | 0 | 0 | 0
  Month 24 | 1.29 (1.854) |  |  |
  Month 30: number analyzed (Participants) | 13 | 0 | 0 | 0
  Month 30 | 1.23 (1.347) |  |  |
  Month 36: number analyzed (Participants) | 14 | 0 | 0 | 0
  Month 36 | 1.46 (1.864) |  |  |
  Month 42: number analyzed (Participants) | 0 | 0 | 0 | 0
  Month 48: number analyzed (Participants) | 6 | 0 | 0 | 0
  Month 48 | 1.28 (2.274) |  |  |

4. Secondary Outcome: Descriptive Statistics of Physician Global Assessment Score
Description: Physician and Patient Global Assessment of disease status was measured by Visual Analogue Scale (VAS) (0-100 mm) for EU patients and Numerical Rating Scale (NRS) (0-10) for Korea patients where higher scores indicated poorer status.
  Descriptive statistics for actual value of Global Assessment Score were summarized by analysis group and every six months including Day 0. For the summary table, each score of Korea patients in NRS was transformed by multiplying 10. Scores are from 0 to 100, with higher scores indicating more disease activity.
Time Frame: Day 0 ~ Month 48 (every 6 months ±6 weeks)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Remsima | Switch to Remsima | Remicade | Switch to Remicade
Number analyzed (Participants) | 98 | 20 | 3 | 4
score on a scale
  Day 0: number analyzed (Participants) | 97 | 20 | 2 | 4
  Day 0 | 54.3 (28.09) | 20.0 (17.17) | 30.0 (14.14) | 22.5 (18.93)
  Month 6: number analyzed (Participants) | 86 | 16 | 3 | 4
  Month 6 | 16.5 (17.19) | 13.1 (7.93) | 6.7 (11.55) | 20.0 (14.14)
  Month 12: number analyzed (Participants) | 55 | 14 | 1 | 2
  Month 12 | 15.6 (16.80) | 11.4 (3.63) | 30.0 | 5.0 (7.07)
  Month 18: number analyzed (Participants) | 28 | 2 | 1 | 0
  Month 18 | 7.8 (8.93) | 30.0 (14.14) | 40.0 |
  Month 24: number analyzed (Participants) | 17 | 0 | 0 | 0
  Month 24 | 2.2 (4.75) |  |  |
  Month 30: number analyzed (Participants) | 13 | 0 | 0 | 0
  Month 30 | 0.9 (0.76) |  |  |
  Month 36: number analyzed (Participants) | 14 | 0 | 0 | 0
  Month 36 | 1.9 (2.63) |  |  |
  Month 42: number analyzed (Participants) | 0 | 0 | 0 | 0
  Month 48: number analyzed (Participants) | 6 | 0 | 0 | 0
  Month 48 | 2.2 (3.87) |  |  |

5. Secondary Outcome: Descriptive Statistics of Patient Global Assessment Score
Description: as for outcome 4
Time Frame: Day 0 ~ Month 48 (every 6 months ±6 weeks)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Remsima | Switch to Remsima | Remicade | Switch to Remicade
Number analyzed (Participants) | 98 | 20 | 3 | 4
score on a scale
  Day 0: number analyzed (Participants) | 97 | 20 | 2 | 4
  Day 0 | 54.0 (30.76) | 25.5 (20.89) | 25.0 (21.21) | 40.0 (29.44)
  Month 6: number analyzed (Participants) | 86 | 16 | 3 | 4
  Month 6 | 21.5 (22.59) | 20.6 (13.89) | 23.3 (25.17) | 35.0 (34.16)
  Month 12: number analyzed (Participants) | 55 | 14 | 1 | 2
  Month 12 | 21.3 (23.52) | 19.3 (15.92) | 30.0 | 40.0 (42.43)
  Month 18: number analyzed (Participants) | 28 | 2 | 1 | 0
  Month 18 | 21.3 (30.37) | 25.0 (7.07) | 30.0 |
  Month 24: number analyzed (Participants) | 17 | 0 | 0 | 0
  Month 24 | 3.1 (4.87) |  |  |
  Month 30: number analyzed (Participants) | 13 | 0 | 0 | 0
  Month 30 | 2.1 (1.38) |  |  |
  Month 36: number analyzed (Participants) | 14 | 0 | 0 | 0
  Month 36 | 2.6 (2.79) |  |  |
  Month 42: number analyzed (Participants) | 0 | 0 | 0 | 0
  Month 48: number analyzed (Participants) | 6 | 0 | 0 | 0
  Month 48 | 2.8 (3.60) |  |  |

6. Secondary Outcome: Descriptive Statistics of Spinal Pain Score
Description: Patient Assessment of Spinal Pain will be measured by VAS (0-100 mm) for EU patients and NRS (0-10) for Korea patients where higher scores indicates more severe pain.
  Descriptive statistics for actual value of Spinal Pain Score will be summarized by analysis group and every six months including Day 0. For the summary table, each score of Korea patients in NRS will be transformed by multiplying 10. Scores are from 0 to 100, with higher scores indicating more pain as assessed by the patient.
Time Frame: Day 0 ~ Month 48 (every 6 months ±6 weeks)
Population: The Efficacy Analysis set consisted of all patients who received at least one infliximab dose (Remsima or Remicade) and providing at least one post treatment efficacy result during the analysis period. This study's primary objective is to compare RemsimaTM in patients with AS with patients receiving other anti-TNF drugs', especially with 'Remicade'. Therefore Switch to Remsima II" and "Switch to Other Anti-TNF" groups' are excluded from the results.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Remsima | Switch to Remsima | Remicade | Switch to Remicade
Number analyzed (Participants) | 98 | 20 | 3 | 4
score on a scale
  Day 0: number analyzed (Participants) | 97 | 20 | 2 | 4
  Day 0 | 52.9 (29.84) | 23.5 (19.81) | 25.0 (21.21) | 42.5 (26.30)
  Month 6: number analyzed (Participants) | 86 | 16 | 3 | 4
  Month 6 | 18.7 (20.83) | 21.9 (16.42) | 6.7 (11.55) | 27.5 (27.54)
  Month 12: number analyzed (Participants) | 55 | 14 | 1 | 2
  Month 12 | 19.8 (22.70) | 22.1 (14.77) | 30.0 | 25.0 (35.36)
  Month 18: number analyzed (Participants) | 28 | 2 | 1 | 0
  Month 18 | 16.3 (26.78) | 15.0 (7.07) | 30.0 |
  Month 24: number analyzed (Participants) | 17 | 0 | 0 | 0
  Month 24 | 3.1 (4.87) |  |  |
  Month 30: number analyzed (Participants) | 13 | 0 | 0 | 0
  Month 30 | 2.0 (1.35) |  |  |
  Month 36: number analyzed (Participants) | 14 | 0 | 0 | 0
  Month 36 | 2.4 (2.79) |  |  |
  Month 42: number analyzed (Participants) | 0 | 0 | 0 | 0
  Month 48: number analyzed (Participants) | 6 | 0 | 0 | 0
  Month 48 | 2.7 (3.72) |  |  |

ADVERSE EVENTS:
Time Frame: Duration of study participation (up to 5 years)
Description: Adverse events were summarized by all analysis groups.
Arm/Group | Remsima | Switch to Remsima I | Switch to Remsima II | Remicade | Switch to Remicade I | Switch to Remicade II | Other Anti-TNF | Switch to Other Anti-TNF
All-Cause Mortality (participants affected / at risk) | 1/124 | 0/23 | 0/10 | 0/3 | 0/5 | 0/0 | 0/146 | 0/18
Serious Adverse Events (participants affected / at risk) | 14/124 | 1/23 | 2/10 | 0/3 | 0/5 | 0/0 | 11/146 | 0/0
Other Adverse Events (participants affected / at risk) | 50/124 | 9/23 | 9/10 | 2/3 | 2/5 | 0/0 | 43/146 | 7/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Remsima (N=124) | Switch to Remsima I (N=23) | Switch to Remsima II (N=10) | Remicade (N=3) | Switch to Remicade I (N=5) | Switch to Remicade II (N=0) | Other Anti-TNF (N=146) | Switch to Other Anti-TNF (N=0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lip oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sudden death (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelocystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tuberculosis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Obsessive-compulsive disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Remsima (N=124) | Switch to Remsima I (N=23) | Switch to Remsima II (N=10) | Remicade (N=3) | Switch to Remicade I (N=5) | Switch to Remicade II (N=0) | Other Anti-TNF (N=146) | Switch to Other Anti-TNF (N=18)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 6 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 12 | 1 | 1 | 0 | 0 | 0 | 12 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 5 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 0 | 3 | 1 | 0 | 0 | 3 | 2
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test Increased (Investigations) | 5 | 1 | 1 | 0 | 0 | 0 | 5 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 1 | 0 | 0 | 0 | 0 | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 4 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Hypertension (Vascular disorders) | 7 | 0 | 0 | 1 | 0 | 0 | 1 | 1
OTORRHOEA (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Uveitis (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transminases increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperlipideamia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2015-06-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT02557308/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/08/NCT02557308/SAP_001.pdf